CLINICAL TRIAL: NCT00186472
Title: Intervention to Decrease Anxiety in Parents of Infants in the Neonatal Intensive Care Unit (NICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Richard Shaw, M.D., Stanford University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIH 5 T 32 MH19908-7
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2006-12

CONDITIONS: Anxiety; Acute Stress Disorder; Posttraumatic Stress Disorder; Depression
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic; Depression

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Treatment

SUMMARY:
Infants born premature face numerous medical problems, causing significant anxiety for their parents. Parents experience a range of negative emotions including concern for the health and well being of their fragile infant, guilt, and disappointment. Research has indicated that having an infant in the Neonatal Intensive Care Unit (NICU) is highly stressful for parents and multiple studies have demonstrated that parents can develop significant psychological reactions to this experience. Specifically, many parents develop clinically significant anxiety disorders such as acute stress disorder (ASD) and posttraumatic stress disorder (PTSD). This not only impacts the mental well-being of the parents, but also can lead to problems with the parent-infant relationship, and, in turn, negatively impact the infant and the family as a whole. Despite the reported negative effects parents experience due to the stress of having an infant on the NICU, surprisingly little research has examined how to reduce parents' symptoms of anxiety. Because parents play an essential role in the care of their infant after discharge from the NICU, treating the parent's emotional distress is highly important. The purpose of this study is to examine the efficacy of a cognitive-behaviorally based intervention in reducing parents' symptoms of anxiety associated with having an infant on the NICU. This treatment is modeled after treatments that have proven effective with parents of children with other types of medical problems, for example, parents of children with cancer. It is the hope of the investigators that this intervention will effectively reduce symptoms of anxiety of NICU parents as well as the likelihood of developing subsequent psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Participants speak either English or Spanish;
3. The participant's infant is expected to live;
4. The participant's infant was born at Lucile Packard Children's Hospital or transferred to the hospital within 72 hours;
5. Participant's infant is over 1000 grams

Exclusion Criteria:

1. Individuals under 18 years of age;
2. Individuals who do not speak either English or Spanish;
3. Individuals whose infant was not born at or transferred to (within 72 hours of The infant's birth) Lucile Packard Children's Hospital;
4. Individuals whose infant has a life threatening condition and is not expected to survive;
5. Current drug abuse/dependence

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Bernard, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States